CLINICAL TRIAL: NCT03320733
Title: Comparison of Volume-Mode 2-Rotation kV-mA Switching Dual Energy Computer Tomography (CT) and of CT Subtraction Imaging With Magnetic Resonance Imaging for the Identification of Enhancing Septa and Mural Nodules in Cystic Pancreatic Lesions
Brief Title: Comparison Between Dual Energy/Subtraction CT With MRI for the Identification of Predictors of Malignancy in Cystic Pancreatic Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 17-5314.0
Record Dates: First submitted 2017-09-19; First posted 2017-10-25 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Pancreatic Cyst
Keywords: dual energy CT
MeSH Terms: conditions — Pancreatic Cyst

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical (Experimental): Includes patients who will undergo surgery for their pancreatic cysts.
  In addition to the routine pre-operative CT abdomen performed for surgical planning purposes, these patients will receive Dual Energy CT scan with subtraction imaging before surgery.
  Interventions: Diagnostic Test: Dual energy CT scan with subtraction imaging
- Surveillance (Experimental): Includes patients who are undergoing surveillance for their pancreatic cysts.
  Dual Energy CT scan with subtraction imaging will be performed in addition to the standard-of-care surveillance method of MRI scans.
  Interventions: Diagnostic Test: Dual energy CT scan with subtraction imaging

INTERVENTIONS:
Diagnostic Test: Dual energy CT scan with subtraction imaging — The single source V2R kmAS dual energy CT system has several theoretical advantages compared, such as perfectly matched X-ray paths and the possibility of performing dual-energy processing using projection data.
  Subtraction imaging is an accurate deformable registration algorithm that allows creation of iodine maps from matched pre- and post-contrast acquisitions. This algorithm can be applied to both single and dual energy CT.

SUMMARY:
Cystic pancreatic lesions are increasingly detected incidentally in imaging studies, reportedly in up to 45% of the abdominal Magnetic Resonance (MR) examinations. The majority of these lesions have potential to become cancer, therefore requiring surgery or imaging follow-up to monitor the development of features indicative of malignant transformation. Abdominal MR is the current standard of care for the follow-up of pancreatic cysts (PCs). However, MR is expensive and access is limited, In our institution, more than 35 MR studies for assessment of PCs were performed each month in 2015, placing a significant burden on the health care system that includes contributing to longer MR wait times for other indications.

The investigators will compare MR to two new computed tomography (CT) techniques - dual energy CT (DECT) and Subtraction imaging - with regards to their ability to detect features associated with increased risk of malignancy (enhancing septa and mural nodules) in PCs. For cases where there is disagreement between these 2 CT techniques and MR, histopathology of the surgical specimen or the results of Endoscopic Ultrasound (EUS) will serve as reference standard.

Using DECT or Subtraction instead of MR for the assessment and follow-up of PCs would save significant healthcare costs and MR slots, which could be released to other indications and to reduce waiting times. Furthermore, if DECT and/or Subtraction imaging end up demonstrating to be superior to MR for this purpose, patients with cystic pancreatic lesions could have a direct benefit.

DETAILED DESCRIPTION:
With the rapid technological advancement, growth and widespread use of cross-sectional imaging, there has been increased detection of pancreatic cystic lesions (PCs). The reported incidence of pancreatic cysts varies widely, with some studies reporting incidental pancreatic cysts detected in 0.7-2.6 % of asymptomatic adults undergoing imaging. The incidence reportedly increases with age with a greater than 8% detection rate in those over age 80 years. The prevalence of a cystic pancreatic lesion in one autopsy series was as high as 24%. For MRI, the frequency of detection of a pancreatic cyst is significantly higher than that of CT, with a reported prevalence of 13-45 % for MRI. Consequently, there has been a significant increased number of MRs ordered for follow-up of these lesions. In our institution, more than 35 MR studies for assessment of PCs were performed each month in 2015. This represents greater than 5% of all abdominal/pelvic MR examinations, and this number appears to be growing. The impact on health care system - particularly on health care costs as well as MR waiting times for patients with other conditions - is significant. For instance, in our institution, the average waiting period in 2015 for an outpatient MR enterography for patients with Crohn's disease is over 6 months.

Recently, dual energy CT (DECT) has proven to be robust and clinically useful for many abdominal applications (including solid pancreatic masses). The investigators expect V2R kVmAS DECT and Subtraction imaging - two promising techniques which have scarcely been investigated in abdominal disease processes in the literature - to prove to be very useful for the characterization of pancreatic cysts and to demonstrate comparable diagnostic accuracy compared to MR

The aim of the study is to investigate whether optimized DECT and/or Subtraction imaging protocols allow for characterization of cystic pancreatic lesions (in particular, the presence of enhancing septa and mural nodules) with a diagnostic accuracy equivalent to or greater than MRI.

This is a prospective, single-institution study in patients who are being evaluated or followed for known pancreatic cystic lesions who are planned for a CT and MRI scan. All MRI scans performed during the study period will be monitored prospectively to identify consecutive patients undergoing MRI for assessment or follow-up of pancreatic cystic lesions and meeting the study inclusion/exclusion criteria.

Patients will be divided into two groups:

- Group 1 includes patients who will undergo surgery for their pancreatic cysts: For these patients, a pre-operative CT abdomen is routinely performed for surgical planning purposes. The treating surgeon will contact the study team to arrange for the CT scan - which will include a DECT scan - to be performed on the appropriate scanner.

- Group 2 includes patients who are undergoing surveillance. For these patients, the standard of care is typically to follow these patients annually with serial MRI scans.

In cases where findings on MRI are in doubt, a CT scan - which will include a DECT scan - will be requested as a problem solving tool and part of the standard of care.

For most patients, a CT scan is not required as part of the standard of care. In these cases, patients will be recruited and consented for an additional CT scan - which will include a DECT scan - to be performed within 6 months of their MRI. This CT scan is in addition to the standard of care. The patient will be recruited at the time of the first follow-up appointment with their treating surgeon after their MRI scan.

ELIGIBILITY:
Inclusion criteria:

* Patients of all ethnic groups older than 40 years old
* Cystic pancreatic lesions larger than 1 cm documented by MR
* Scheduled for surgery (Group 1) or undergoing surveillance (Group 2) for a pancreatic cyst by a hepatobiliary surgeon at UHN (University Health Network)

Exclusion criteria:

* Patients with contraindication for contrast-enhanced CT or MRI
* Pregnancy
* Patients who do not consent to the study
* Patients younger than 40 years old or with pancreatic cysts less than 1 cm

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity | 2 years
  Sensitivity of Dual Energy CT in prediction of malignancy for pancreatic cysts > 1cm.
Specificity | 2 years
  Specificity of Dual Energy CT in prediction of malignancy for pancreatic cysts > 1cm.
Positive predicative value | 2 years
  Positive predicative value (PPV) of Dual Energy CT in prediction of malignancy for pancreatic cysts > 1cm.
Negative predicative value | 2 years
  Negative predicative value (NPV) of Dual Energy CT in prediction of malignancy for pancreatic cysts > 1cm.

SECONDARY OUTCOMES:
Parameters optimization HU | 2 years
  Cutoffs of Hounsfield Units (HU) on Subtraction imaging for true enhancing components of pancreatic cysts.
Parameters optimization keV | 2 years
  Optimal keV value on virtual monochromatic DECT images for true enhancing components of pancreatic cysts.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Guimaraes, MD, Principal Investigator — University of Toronto, Department of Medical Imaging
Locations (1):
- University of Toronto, Department of Medical Imaging, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No